CLINICAL TRIAL: NCT06253299
Title: How Applying Cold to Different Side Neck Region Affects Venous Cannulation Pain: Prospective Randomized Controlled Study
Brief Title: Effect of Cold Application to Different Side Neck Region on Venous Cannulation Pain
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Senay Canikli, medical specialist (Anesthesiology and Reanimation), Samsun University
Other Study IDs: GOKAEK 2024/3/9
Record Dates: First submitted 2024-02-01; First posted 2024-02-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Venous Canulation Pain; Nervous Vagus; Left Side; Right Side

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group L: Just before the vascular access is opened, a 4x5 cm sized marble stone will be applied to the carotid in the left lateral neck region (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SKM)) for 30 seconds, and then the vascular access will be opened
  Interventions: Other: marble stone
- Group R: Just before the vascular access is opened, a 4x5 cm cold marble stone will be held on the carotid in the right lateral neck area (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SKM)) for 30 seconds (sec), and then the vascular access will be opened.
  Interventions: Other: marble stone

INTERVENTIONS:
Other: marble stone — Marble stones with dimensions of 4x5 cm will be used for cold application. When placed in the freezer compartment of the refrigerator at -10°C (Celsius) for 4 minutes, they cool down to 11°C. Subsequently, in 1 minute, the temperature rises to 12°C when held in the palm. "After being placed on a table at room temperature, it reaches 18°C in 5 minutes."

SUMMARY:
Intravenous (iv) cannulation is one of the most common applications performed by anesthesiologists in and outside the operating room. It is necessary to provide vascular access before any anesthetic procedure. Venous cannulation is a moderately painful procedure and is uncomfortable for patients, and the pain of intravenous cannulation may increase the patient's stress. Various methods are used to reduce cannulation pain. Stimulation of the N. Vagus is also among these methods (1). The branches of N. Vagus are densely located under the skin in the auricle and on the lateral aspect of the neck. It is thought that the dominance of the right and left vagal nerve over different systems is different. For example; While the right vagal branches are thought to be more effective on heart rate, the left side vagal branches are thought to be more effective in the treatment of refractory epilepsy. Purpose: Our aim in this study is to evaluate the vascular access pain in our patients to whom investigator applied venous cannulation from the back of the hand before anesthesia, by stimulating the Vagus Nerve with cold application to the neck area on both sides separately.

DETAILED DESCRIPTION:
Various methods are being tried to reduce cannulation pain. Methods such as injection of local anesthetic into the intervention area, use of topical anesthetic, application of ice, and vibrating buzz application have been used to relieve the patient's pain and distract him. There are many different methods of stimulating the vagus nerve. Valsalva maneuver is a mechanism that stimulates Nervus Vagus (N. Vagus). Stimulation of the vagus nerve is thought to have an analgesic effect (2). Stimulation of the vagal nerve has an antinociceptive effect by triggering the baroreceptor reflex arc. It is thought that antinociceptive substance P-like substance is released with the activation of the baroreceptor reflex arc. The areas where N. Vagus is most superficial in the periphery are inside the auricle and the lateral neck region. It is also known that cold application to the lateral neck area reduces the heart rate by stimulating the N. Vagus (5). The degree of effect of vagal stimulation from different sides on different systems may be different (2,3). Applying cold to the neck area will have an antinociceptive effect by activating the baroreceptor reflex arc by stimulating the N. Vagus, and the degree of this effect may be effective differently with stimulation from the right or left side.

Method:

Patients aged 18-75 who will undergo elective surgery (except those who will undergo oncological surgery and those who will undergo cesarean section) will be included in the study. These patients will be evaluated at the anesthesia clinic before the operation. Those who have a scar on the back of the hand, who have had surgery on the back of the hand, who have psoriasis, who have peripheral vascular disease, who use chronic analgesics, who use opioids, who use steroids, who use gabapentinoids, who have a history of substance use, who have peripheral neuropathy, who have received oncological treatment and who have limited cooperation. patients will not be included in the study. Power analysis was done with G*Power 3.1.9.7 program. Before the study, the program was run to calculate the sample size to be equally distributed among the groups, assuming α = 0.05, power (1-β) = 0.80, effect size = 0.5. According to this program, the total number of samples is 128 and there are 64 people in each group. Taking into account recording errors, 70 people in each group and the total sample size was determined as 140 people) will be randomized into 2 groups: Group R (right side) and Group L (left side). The lottery method will be used for randomization.

Group R: Just before the vascular access is opened, a 4x5 cm cold marble stone will be held on the carotid in the right lateral neck area (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SKM)) for 30 seconds (sec), and then the vascular access will be opened.

Group L: Just before the vascular access is opened, a 4x5 cm sized marble stone will be applied to the carotid in the left lateral neck region (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SKM)) for 30 seconds, and then the vascular access will be opened.

Before vascular access is established, heart rate (HR), respiratory rate (RR) and noninvasive blood pressure (NIBB) will be recorded. HR, RR and NIBB values will be recorded after application to the neck area. Then, an 18-gauge (green colored) intraket will be inserted one time by the same experienced practitioner on the back of the left hand, and the patients will be asked to rate their pain levels between 0-10 according to the NRS and this value will be recorded. HR, RR and NIBB values will also be recorded. Patients who cannot be cannulated at once will be excluded from the study.

Patients' data will be recorded using SPSS 18 program. The relationship between the NRS scores of both groups and the patients' HR, RR and NIBB values before cold application, after cold application and during vascular access will be evaluated. Descriptive statistics, analysis of variance and chi-square test will be used to evaluate the data. Mean±standard deviation and percentages will be used in descriptive statistics. Results will be evaluated at 95% confidence interval and significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA I,II,III patients
* Patients who will undergo elective surgery

Exclusion Criteria:

* -Patients undergoing emergency surgery
* Patients who will undergo oncological surgery
* Pregnant patients
* Patients with scars on the back of the hand
* Who had surgery on the back of the hand
* Patients with psoriasis
* Those with peripheral vascular disease
* Patients using chronic analgesics
* Patients using opioids
* Those who use steroids
* Those who use gabapentinoids
* Those with a history of substance use
* Those with peripheral neuropathy
* Patients who have received oncological treatment
* Patients with limited cooperation
* Patients using medications that affect heart rate (such as beta blockers, calcium channel blockers)
* Patients with rhythm disorders
* Patients using cardiac pacemaker

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-75 who will undergo elective surgery
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Venous cannulation pain | preoperative period
  Venous cannulation pain will be evaluated with the numerical pain scale (NRS).

SECONDARY OUTCOMES:
heart rate | preoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Senay canikli adıgüzel, Principal Investigator — Samsun University
Locations (1):
- Şenay Canikli Adıgüzel, Ataşehir, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://dx.doi.org/10.4097/kjae.2016.69.1.27